CLINICAL TRIAL: NCT04464057
Title: Safety and Effectiveness of Early Feeding After Bowel Anastomosis in Neonates or Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weibing Tang (Other)
Responsible Party: Sponsor-Investigator, Weibing Tang, Chief of neonatal surgery department of Nanjing Children's Hospital, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NanjingCH
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Enteral Feeding; Neonate; Infant; Intestinal Anastomosis Complication
Keywords: oral feeding; early enteral nurtrion; Intestinal anastomosis; neonate; infant

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized controlled clinical study. A total of 285 inpatients (95 experimental groups and 190 control groups) were enrolled to evaluate the safety and effectiveness of early feeding in neonates and infants after intestinal anastomosis
Who Masked: Participant
Masking Description: According to age and disease, the first pairing design, three pairs (experimental group: control group = 1:2), after pairing three subjects randomly assigned to the experimental group, the other two to the control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The patients in the experimental group would be given early oral feeding within 24-48 hours after intestinal anastomosis. Start taking it at 24-48 hours after surgery until discharged. The initial dose is 1ml/kg.h, which is gradually increased to 100ml/kg daily.
  Interventions: Dietary Supplement: early oral feeding or early enteral nurtrion
- control group (No Intervention): The control group would be given early oral feeding within 4-5 days after intestinal anastomosis. Start taking it at 4-5 days after surgery until discharged. The initial dose is 1ml/kg.h, which is gradually increased to 100ml/kg daily.

INTERVENTIONS:
Dietary Supplement: early oral feeding or early enteral nurtrion — The patients in the experimental group were fed orally within 24-48 hours after intestinal anastomosis. Start taking it at 24-48 hours after surgery until discharged. The initial dose is 1ml/kg.h, which is gradually increased to 100ml/kg daily.
  Arms: experimental group

SUMMARY:
The study is primary designed to evaluate the safety and effectiveness of early feeding after bowel anastomosis, and observe the effect of early postoperative feeding on promoting postoperative rehabilitation and reducing parenteral nutrition

DETAILED DESCRIPTION:
Intestinal anastomosis is a common operation for the treatment of digestive tract diseases of newborns and infants. It is not be defined that when should begin oral feeding after intestinal anastomosis. Poor anastomotic healing or anastomotic leakage is the most serious complication after intestinal anastomosis, which often leads to severe abdominal infection, peritonitis and even death. Nowadays, it is believed that the causes of poor anastomotic healing or anastomotic leakage are various, including contaminated during the operation, the blood supplyment of the bowel edges at both ends of the anastomosis, anemia, anastomosis technique, type of surgery (selective or emergency), and anastomotic tension . The traditional view is that early feeding may increase the anastomotic tension, which may lead to poor anastomotic healing or leakage, so a lot of surgeons often take a fasting for 4-5 days after intestinal anastomosis to ensure good anastomotic healing, however there is no enough evidence for this view. On the contrary, the current research confirms that after intestinal anastomosis, under fasting conditions, the digestive system still has 1-2 liters of fluid through the anastomosis, so even if it is given postoperative oral feeding, It would not excessively increase the digestive fluid through the anastomosis. Obviously, the early guess that the anastomotic tension is increased is lacking in theoretical evidence. In recent years, with the in-depth study of intestinal function, intestinal mucosal barrier function and intestinal flora, early enteral nutrition has stretched more and more attention, which is believed could stimulate intestinal digestive fluid secretion, promote intestinal mucosal metabolism and repair, avoid intestinal villi atrophy, reduce intestinal bacterial translocation, promote intestinal function recovery and intestinal peristalsis. Postoperative intestinal obstruction is also an important reason for hindering early enteral nutrition, but current research believes that postoperative intestinal obstruction is often temporary, and in most cases will be relieved 4-8 hours after surgery. European Society of Parenteral Enteral Nutrition (ESPEN ) recommended that enteral nutrition should be performed within 24 hours after intestinal anastomosis, but it needs to be fully evaluated according to the children's own tolerance and the type of surgery. A large number of studies and meta-analysis have confirmed that early enteral nutrition is safe and feasible after intestinal anastomosis in adults, but there are still few studies in children, especially whether early enteral surgery can be performed after intestinal anastomosis is currently rarely reported in neonates and infants. This study evaluated the feasibility and effectiveness of early oral enteral nutrition in neonates and infants after intestinal anastomosis through a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* (1)neonates or infants less than 12 months (2)Intestinal anastomosis, including small intestine and colon anastomosis

Exclusion Criteria:

* (1) Premature infants or children with a weight of less than 2.5 kg during surgery are excluded (2) Exclude cases of severe abdominal infection (3) Exclude cases of severe imbalance of the proximal and distal intestinal canal of the anastomosis (such as intestinal atresia)

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 947 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage or poor anastomotic healing | 1-7days after early oral feeding
  Feces flow out from the site of the anastomosis into the abdominal cavity
Gastrointestinal symptoms:nausea, vomiting, diarrhea, abdominal pain and abdominal distent. | 1-14days after early oral feeding
  There may be some unexpected symptoms happen after early oral feeding after anastomosis such as Nausea, vomiting, diarrhea, abdominal pain and abdominal distent.
indexs of stress:C-reactive protein, interleukin 6, cortisol | The first day and third day after early oral feeding
  Some indexs could be defined as indicators of the severity of the stress response
indexs of nurtrion:weight, serum albiumin,serum prealbumin and serum retinol binding protein | The seventh day after anastomosis
  Some indexs could be defined as indicators of the nutriton status

SECONDARY OUTCOMES:
indexs of recovery after surgery:Time to first bowel movement, time to use intravenous nutrition and total postoperative hospital stay | 1-14 days after surgery.
  Some indexs could be defined as indicators of recovery after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Tang, Dr, Study Director — Children's Hospital of Nanjing Medical University
Locations (2):
- China (2):
  - Anhui Provincial Children's Hispital, Hefei, Anhui
  - Xuzhou CHildren's Hospital Affilated to Xuzhou Medical College, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No
The data of the study would be shared with othe researchers.

REFERENCES:
- [Derived] Lu C, Sun X, Geng Q, Tang W. Early oral feeding following intestinal anastomosis surgery in infants: a multicenter real world study. Front Nutr. 2023 Jul 20;10:1185876. doi: 10.3389/fnut.2023.1185876. eCollection 2023. PMID 37545580

DOCUMENTS (1):
  • Study Protocol (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT04464057/Prot_000.pdf